CLINICAL TRIAL: NCT06047249
Title: Study on the Mechanism of Prevotella Copri Promoting the Occurrence and Development of Atherosclerosis
Acronym: SOMOFPcopri
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hai Tian (Other)
Responsible Party: Sponsor-Investigator, Hai Tian, Clinical Professor, The Second Affiliated Hospital of Harbin Medical University
Organization: The Second Affiliated Hospital of Harbin Medical University (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2ndHarbinMU2022
Record Dates: First submitted 2023-07-17; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Coronary heart disease group (No Intervention): 16SrDNA sequencing and ELISA test were carried out for patients over 50 years old who reported coronary atherosclerosis after coronary angiography or coronary angiography with CT examination to detect the abundance of Prevotella in their intestines, the concentration of 5-hydroxytryptamine, branched chain amino acids and lipopolysaccharide in their blood
- Non coronary heart disease group (No Intervention): For patients over 50 years old who reported no coronary atherosclerosis after coronary angiography or CTA examination, 16SrDNA sequencing and ELISA tests were carried out to detect the abundance of Prevotella in the intestinal tract, the concentration of 5-hydroxytryptamine, branched chain amino acids and lipopolysaccharide in the blood
- KAP group (Experimental): Conduct a survey on the relationship between coronary heart disease and dietary patterns among hospitalized patients in the form of KAP Popular Science Research. After the survey, conduct scientific popularization of relevant knowledge, conduct a satisfaction questionnaire survey after surgery, and collect data on preoperative and postoperative examinations and laboratory tests
  Interventions: Behavioral: KAP Popular Science Research
- Non KAP group (Sham Comparator): Investigators will not conduct a survey on the relationship between coronary heart disease and dietary patterns among hospitalized patients, conduct science popularization, and conduct a satisfaction questionnaire survey after surgery
  Interventions: Behavioral: No KAP Popular Science Research

INTERVENTIONS:
Behavioral: KAP Popular Science Research — By conducting a survey questionnaire, investigate the knowledge, attitude, and practice tendencies of patients and their caregivers towards a certain disease, and conduct relevant science popularization；Pre discharge satisfaction survey questionnaire
  Arms: KAP group
Behavioral: No KAP Popular Science Research — Pre discharge satisfaction survey questionnaire
  Arms: Non KAP group

SUMMARY:
Mainly studying the correlation between the abundance of Prevotella copri （P.copri） in the gut microbiome and the progression of clinical coronary atherosclerotic heart disease（CAD） patients, and confirming that an increase in P.copri abundance will accelerate the occurrence and development of CAD disease, accompanied by an increase in serum Branched chain amino acid（BCAA）, lipopolysaccharide（LPS）, and serotonin; For people who mainly consume a high carbon water diet, blood sugar is a stronger risk factor for AS compared to blood lipids; Explore the KAP status（Study composes of Knowledge, attitude, and practice） of coronary heart disease patients and their caregivers regarding coronary heart disease and diet, and investigate whether the popularization of science after KAP investigation can change the treatment effect of patients.

DETAILED DESCRIPTION:
Confirming the progression of coronary heart disease in patients and the proportion of P.copri in the gut microbiome; Confirming that due to the increased abundance of P.copri, factors related to blood glucose metabolism disorders are more associated with the progression of CAD disease compared to lipid factors; Confirming that P.copri induces insulin resistance and inflammation in the body while altering intestinal permeability through the synthesis of BCAA, LPS, and serotonin;; Through controlled experiments conducted at our center, investigators effectively popularized disease science to patients and their caregivers, promoted their participation in disease treatment, and confirmed that the KAP survey method can optimize patient treatment effectiveness, improve doctor-patient relationships, and enhance patient hospitalization experience. Through this research project, investigators explore the application of KAP research in the form of a questionnaire in this discipline. Through KAP research, investigators aim to popularize knowledge about dietary patterns and coronary heart disease among multi center coronary heart disease patients and their caregivers. investigators also investigate the "knowledge", "belief", and "behavior" of current coronary heart disease patients and their caregivers regarding coronary heart disease diagnosis and treatment knowledge, and conduct a knowledge lecture, Establish a new model for mastering, attitudes, and actions related to the diagnosis and treatment of coronary heart disease among patients and their accompanying caregivers through data push and other forms, while also providing theoretical and practical basis for subsequent related research. Through this project, investigators will discuss the feasibility of KAP survey in increasing patients' subjective initiative, improving doctor-patient relationships, and promoting the effectiveness of patient treatment. investigators will also discuss its promotion and inclusion in routine diagnostic and treatment methods.

ELIGIBILITY:
Inclusion Criteria:

1. Atherosclerosis mechanism research: diagnosis is made through clinical diagnostic technical indicators, mainly coronary CT or coronary angiography. Experimental group: patients with coronary heart disease are identified; Control group: Admitted patients without coronary heart disease but may have other heart diseases or risk factors; Age:>50 years old
2. KAP Study: Coronary Heart Disease Patients and Their Families

Exclusion Criteria:

1. Atherosclerosis mechanism research: age<50 years old; Patients with a history of coronary heart disease or surgery; Patients with systemic diseases, including liver and kidney diseases (with serum creatinine levels>2mg/dL (176.8 μ Mol/dL), collagen diseases, etc; Patients who have been using antibiotics within the past 6 months; Patients with malignant tumor disease
2. KAP Study: Non coronary heart disease patients and their caregivers

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-07-07 (Estimated); Study Completion 2024-07-07 (Estimated)

PRIMARY OUTCOMES:
Concentration of Brain Natriuretic Peptide | Within 7 days after surgery
  Blood sampling and testing
Concentration of myocardial enzyme | Within 7 days after surgery
  Blood sampling and testing
Concentration of troponin | Within 7 days after surgery
  Blood sampling and testing
questionnaire1 | Within 7 days after admission
  KAP scale，This questionnaire consists of a total of 25 questions, with the first 7 questions being the baseline survey of the subjects, which facilitates statistical information without involving scores. The remaining questions consist of 10 knowledge questions (each desired response was scored 1, maximum K-score was 10), 5 attitude questions (each desired response was scored 1, maximum A-score was 5), and 3 practice questions (this question consists of 5 options, depending on frequency or severity, 1 is obtained when selecting 1 or 2 options, 2 is obtained when selecting 3 options, 3 is obtained when selecting 4 or 5 options, and 5 is obtained when selecting maximum P-score was 5)，higher scores mean a better outcome
questionnaire2 | Within 7 days after surgery
  Composed of 5 questions, choose the expected answer and add 1 point. The higher the score, the better
Prevotella copri abundance | through study completion, an average of 1 year
  16S ribosomal DNA identification sequencing of feces
Concentration of branched chain amino acids | through study completion, an average of 1 year
  Blood sampling and testing
Concentration of serotonin | through study completion, an average of 1 year
  Blood sampling and testing
lipopolysaccharides | through study completion, an average of 1 year
  Blood sampling and testing
Concentration of blood glucose | through study completion, an average of 1 year
  Blood sampling and testing
Concentration of lipids | through study completion, an average of 1 year
  Blood sampling and testing
cardiac ejection fraction | Within 7 days after surgery
  Ultrasonic instrument exploration
cardiac ejection fraction | 7 days before surgery
  Ultrasonic instrument exploration
ejection volume | 7 days before surgery
  Ultrasonic instrument exploration
ejection volume | Within 7 days after surgery
  Ultrasonic instrument exploration
left ventricular size | Within 7 days after surgery
  Ultrasonic instrument exploration
left ventricular size | 7 days before surgery
  Ultrasonic instrument exploration
end diastolic diameter | 7 days before surgery
  Ultrasonic instrument exploration
end diastolic diameter | Within 7 days after surgery
  Ultrasonic instrument exploration
left ventricular end systolic diameter | Within 7 days after surgery
  Ultrasonic instrument exploration
left ventricular end systolic diameter | 7 days before surgery
  Ultrasonic instrument exploration
pulmonary artery pressure | 7 days before surgery
  Ultrasonic instrument exploration
pulmonary artery pressure | Within 7 days after surgery
  Ultrasonic instrument exploration

CONTACTS AND LOCATIONS:
Overall Officials: Hai Tian, Principal Investigator — Harbin Medical University Second Affiliated Hospital
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No